CLINICAL TRIAL: NCT05006937
Title: Prospective, Randomized Study to Assess Patient Satisfaction and Stone Free Effect of High Powered Stone Dusting vs. Fragmentation and Basketing at Time of Ureteroscopy
Brief Title: High Powered Stone Dusting vs. Fragmentation and Basketing at Time of Ureteroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amy Krambeck, Professor of Urology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00214998
Record Dates: First submitted 2021-08-06; First posted 2021-08-16 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Kidney Stone; Ureteral Stone
MeSH Terms: conditions — Kidney Calculi; Ureterolithiasis | interventions — Dust

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- laser dusting (Active Comparator): In the "dusting" arm, the ureteroscope will be advanced into the kidney or ureter over an access wire without an access sheath in place. The identified stone will be dusted using a 200 micron Moses laser fiber at a setting of 0.3-0.6 J and 50-120 Hz using the Moses 2.0 laser system. Stone dusting will continue until the surgeon feels the fragments are all negligible in size and would be able to pass. One small piece will be extracted for analysis and the remainder will be left to pass spontaneously. If there is no evidence of injury or swelling of the ureter at the conclusion of the case a stent will be omitted.
  Interventions: Procedure: Dusting
- basketing (Active Comparator): In the Basketing arm, a ureteral access sheath (UAS) will be placed per standard fashion. The ureteroscope will be introduced into the kidney and the stone fragmented at a setting of 0.8-1.0 J and 6-15 Hz. The resultant fragments will be basket extracted through the sheath for analysis. All fragments will be removed until no residual stone remains. At the time of UAS removal the ureter will be inspected. If there is no evidence of ureteral injury or swelling then a stent will be omitted.
  Interventions: Procedure: Basket extraction

INTERVENTIONS:
Procedure: Dusting — Dusting is when a laser is used to break a stone down into tiny fragments that are able to pass through the urine.
  Arms: laser dusting
Procedure: Basket extraction — Basket extraction is when a small wire basket is used to remove stone fragments.
  Arms: basketing

SUMMARY:
The purpose of this study is to determine the differences in stone free results, patient side effects, and patient satisfaction between dusting vs. basket extraction for kidney and ureteral stones (a kidney stone located in the tube between the kidney and bladder) 6 mm and greater in size undergoing ureteroscopic treatment.

Dusting is when a laser is used to break a stone down into tiny fragments that are able to pass through the urine. Basket extraction is when a small wire basket is used to remove stone fragments.

DETAILED DESCRIPTION:
On the day of surgery, the treatment assigned to the patient will be determined by chance, like flipping a coin. Neither the patient nor the study doctor will choose the treatment type. Each patient will have an equal chance of being given either surgical treatment. One group will have stones treated with high-powered laser dusting and the dust produced will pass spontaneously through the urine. The other group will have stones treated with low power laser fragmentation and stones will be removed using a basket. The surgical procedure will not differ from the treatment a patient would receive if he/she were not in this study.

After surgery, participants will complete a pain assessment questionnaire in the outpatient recovery area before being discharged to go home. Participants will also receive a daily email or text message to assess pain and daily activities. Participants will answer these questions daily until pain has resolved and daily activities have returned to baseline levels.

Six weeks after surgery, participants will undergo an ultrasound to assess for swelling of a kidney due to a build-up of urine (called hydronephrosis), which is standard of practice after ureteroscopy. Participants will also return to the urology clinic 12 weeks after surgery for a standard of care follow up visit. At this visit, participants will undergo standard of care procedures known as renal bladder ultrasound and kidney ureter bladder abdominal x-ray to evaluate for stones. Participants will also complete another pain assessment questionnaire at this appointment.

Researchers will review the medical record to evaluate the effectiveness of the surgery at removing kidney stones and preventing kidney stone recurrence as well as to track quality of life outcomes.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* undergoing ureteroscopic stone extraction
* Stone size 6mm stones or greater and the location to mid ureter or higher
* Willing to sign informed consent form
* Able to read, understand, and complete patient questionnaires, and pain questionnaires

Exclusion Criteria:

* < 18 years of age
* Inability to provide informed consent
* Concomitant surgery (i.e. Percutaneous nephrolithotomy, Holmium laser enucleation of the prostate
* Solitary kidney
* Nephrocalcinosis
* Members of vulnerable patient populations
* Patients without access to a phone that can receive txt messages

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Stone free rate: clinical | 6 weeks
  patients with no clinical evidence of kidney stones on the treated side
Stone free rate: imaging | 6 weeks
  patients with no radiographic evidence of kidney stones on the treated side

SECONDARY OUTCOMES:
Patient quality of life- pain intensity | 12 weeks
  patient quality of life measures as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire Pain Intensity - Short Form 3a. Higher score indicates higher pain levels. Lowest score 3, highest score 15.
Patient quality of life- pain interference | 12 weeks
  patient quality of life measures as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire Pain Interference - Short Form 6b. Higher scores indicate higher levels of pain interference. Lowest score is 6, highest score is 30.
Return to work | 12 weeks
  Days missed from work after surgery
Daily activity level | 12 weeks
  Days until patients have returned to baseline pre-surgery daily activity level

CONTACTS AND LOCATIONS:
Overall Officials: Amy Krambeck, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No